CLINICAL TRIAL: NCT05290532
Title: Effect of Multimodal Postoperative Rehabilitation on Functional and Cognitive Decline, in Elderly Patients Undergoing Urgent Abdominal Surgery: A Randomized Clinical Trial
Brief Title: Effect of Multimodal Postoperative Rehabilitation on Functional and Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital of Navarra (Other)
Collaborators: Fundacion Miguel Servet (Other)
Responsible Party: Principal Investigator, IRENE ESQUIROZ, Principal Investigator, Hospital of Navarra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hospital de Navarra
Record Dates: First submitted 2022-02-10; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Surgery--Complications
Keywords: Elderly patients; Exercises; Cognitive Dysfunction; Quality of life
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial,patient who meet the inclusion criteria will be randomly assigned to the intervention or control group
Who Masked: Investigator
Masking Description: The study participants will be randomized ( ww. randomizer.org) into an intervention group and a control group. the assessment staff will be blinded to the participant randomization assignment, as well as to the main study design ant to what changes we expect to occur in the study outcomes in either group.
  It will not be possible to conceal the group assignment from the staff involved in the training of the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized exercise training (Other): Exercise training. Individual program training 2 days per week during 4 week, after one week of discharge
  Interventions: Other: Individualized exercise training
- No Intervention: Control (No Intervention): Usual care including rehabilitation when necessary

INTERVENTIONS:
Other: Individualized exercise training — The intervention will consist of a multicomponent exercise training program, which will composed of supervised progressive resistance exercise training, aerobic and anaerobic exercises. This training period consist on 2 training sessions of 40 minutes (Warm up 5´+ aerobic exercise 15´+ anaerobic exercise 15´+ stretching 5´)per week during 4 weeks after one week of discharge
  Arms: Individualized exercise training

SUMMARY:
Older adults, especially those with frailty, have a higher risk for complications, functional and cognitive decline after urgent surgery.

These patients have their functional and physiological reserve reduced which makes them more vulnerable to the effects of being bedridden. The consequences are at multiple levels emphasizing the functional loss or cognitive impairment, longer stays, mortality and institutionalization, delirium, poor quality of life and increased use of resources related to health. Exercise training can prevent functional and cognitive decline and modify even the posterior trajectory

DETAILED DESCRIPTION:
This study is a randomized clinical trial conducted in the Department of Surgery of a tertiary public hospital. Patients undergoing urgent abdominal surgery who meet inclusion criteria will be randomly assigned to the intervention or control group. A total of 218 elderly patients undergoing urgent abdominal surgery( control group=109 and intervention group 109) randomly assigned to the intervention or control group.

Patient recruitment will begin in the 4-day after the surgical procedure, which will be identified through the list of patients admitted to the hospital and assigned to the Department. The doctor who decides the inclusion in the intervention or control group will not be the attending physician. Patients or their families (if the patient has cognitive impairment) will be informed of the random inclusion in one group, but will not be informed as to which they belong. Randomization will be performed by applying http://www.randomizer.org/. The information in both the intervention group and the control group will obtained in four different stages: the initial visit and at months 1, 3 and 6 after hospital discharge.

The intervention will consist of a multicomponent exercise training program, which will composed of supervised progressive resistance exercise training, aerobic and anaerobic exercises. This training period consist on 2 training sessions per week during 4 weeks after one week of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older
* Able to tolerate exercise
* Able to ambulate, with or without personal / technical assistance or move unassisted in a wheelchair
* Able to communicate
* Undergoing urgent abdominal surgery
* Barthel Index>60
* Informed consent: must be capable and willing to provide consent

Exclusion Criteria:

* Severe dementia (GDS 7)
* Duration of hospitalization <4 days
* Unwillingness to either complete the study requirements or to be randomized into control or intervention group
* Unstable cardiovascular disease or other unstable medical condition
* Terminal illness
* Myocardial infarction in the past 3 months
* Upper or lower extremity fracture in the past 3 months
* Evisceration

Ages: 70 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in functional capacity of patients | 1, 3 and 6 months after hospitalization discharge
  The functional capacity of patients will be evaluated by the Short Physical Performance Battery (SPPB), which evaluates, balance, gait ability, and leg strength using a single tool. The total score will range from 0 (worst) to 12 points (best).
Changes in Cognitive capacity of patients | 1, 3 and 6 months after hospitalization discharge
  The cognitive-affective status will be measured in the follow up using the Mini Mental State Examination.nThis examination is composed of seven categories designed to assess specific cognitive functions: orientation to time (5 points), orientation to place (5 points), registration of three words (3 points), attention and calculation (5 points), recalling the three words (3 points), language (8 points) and constructive visual capacity (1 point). The MMSE score ranges from zero to 30 points, and lower values indicate possible cognitive deficit
Changes in Quality of life | 1, 3 and 6 months after hospitalization discharge
  Changes in Quality of life will be evaluated by European Quality of Life-5 Dimensions (EuroQol- 5D).
  European Quality of Life-5 Dimensions: comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels, the score will range from 5 (wort) to 15 (best).
Changes in Visual Analogue Scale | 1, 3 and 6 months after hospitalization discharge
  Changes in Visual Analogue Scale (VAS). The VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (100 points) and 'The worst health you can imagine'(0 points).

SECONDARY OUTCOMES:
Postoperative complications | 30 and 90-day
  Comprehensive Complication Index
Length of stay | from the date of admission until the date of discharge
  Length of stay
Mortality | 30 and 90-day
  postoperative mortality
Delirium | from the date of admission until the date of discharge
  Confusion Assessment Method (CAM) The CAM short form assesses four features: 1. acute onset or fluctuating course, 2. inattention, 3. disorganized thinking, and 4. altered level of consciousness. For the diagnosis of delirium, the first two criteria and at least one of the last two are necessary.
Cost per quality-adjusted life year | 6 months post-discharge
  Both direct and indirect study participant costs

CONTACTS AND LOCATIONS:
Overall Officials: IRENE ESQUIROZ, MBBS, Principal Investigator — Hospital of Navarra

REFERENCES:
- [Derived] Esquiroz Lizaur I, Zambom-Ferraresi F, Zambom-Ferraresi F, Ollo-Martinez I, De la Casa-Marin A, Martinez-Velilla N, Recreo Baquedano A, Galbete Jimenez A, Gonzalez Alvarez G, Yarnoz Irazabal MC, Eguaras Cordoba I. Postoperative physical rehabilitation in the elderly patient after emergency surgery. Influence on functional, cognitive and quality of live recovery: study protocol for a randomized clinical trial. Trials. 2024 Sep 4;25(1):584. doi: 10.1186/s13063-024-08406-0. PMID 39232792